CLINICAL TRIAL: NCT04650997
Title: The Mechanical,Physiological and Therapeutic Effects of Eccentric Exercise Combined With Extracorporeal Shockwave Therapy in Athletes With Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSEARS20110215003
Record Dates: First submitted 2020-07-30; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2011-02

CONDITIONS: Patellar Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined (Experimental): 12 weeks eccentric exercise combined with 6 sessions of extracorporeal shockwave therapy in the initial 6 weeks
  Interventions: Behavioral: Eccentric exercise
- Exercise (Sham Comparator): 12 weeks eccentric exercise combined with 6 sessions of sham extracorporeal shockwave therapy in the initial 6 weeks
  Interventions: Behavioral: Eccentric exercise

INTERVENTIONS:
Behavioral: Eccentric exercise — Knee eccentric exercise with sham or focused extrocorporeal shockwave therapy for 12 weeks
  Other Names: Extracoporeal shockwave therapy (Minilith SL1, Storz Medical)

SUMMARY:
Patellar tendinopathy is one of the most common injuries in jumping athletes. Changes in mechanical and physiological properties of tendon are the two proposed forms of pathogenesis. The efficacy of eccentric exercise when applied alone and combined with extrocoporeal shockwave therapy had been reported; however, the underlying treatment mechanisms of pain and dysfunction are not clear. This project aimed to explore the mechanical, physiological and therapeutic effects of eccentric exercise when applied as a single treatment and as an adjunct to extracorporeal shockwave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Competitive athletes
* Pain at the inferior pole of the patella with training for at least 3 months
* Tenderness at the inferior pole of the patella on palpation

Exclusion Criteria:

* Patellofemoral pain syndrome, fat pad irritations, meniscus injury, osteoarthritis, rheumatoid arthritis or infections
* History of fracture over lower limbs and inflammatory myopathies
* Cortisone injuection and other interventions within 3 months
* Contraindication to extracorporeal shockwave therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2014-01-01 (Actual)

PRIMARY OUTCOMES:
Tendon stress in pascals at baseline | Before intervention
  Tendon stress measured by ultrasonography and dynamometry
Change of tendon stress in pascals at 12 weeks | 12 weeks
  Tendon stress measured by ultrasonography and dynamometry
Change of tendon stress in pascals at 16 weeks | 16 weeks
  Tendon stress measured by ultrasonography and dynamometry
Tendon vascularity index as percentage at baseline | Before intervention
  Tendon vascularity measured by power doppler ultrasonography
Change of tendon vascularity index as percentage at 12 weeks | 12 weeks
  Tendon vascularity measured by power doppler ultrasonography
Change of tendon vascularity index as percentage at 16 weeks | 16 weeks
  Tendon vascularity measured by power doppler ultrasonography

SECONDARY OUTCOMES:
Tendon related pain on visual analogy scale at baseline | Before intervention
  Maximal intensity of self-perceived pain in the past 7 days, pain during single-leg declined-squat test
Change of tendon related pain on visual analogy scale at 12 weeks | 12 weeks
  Maximal intensity of self-perceived pain in the past 7 days, pain during single-leg declined-squat test
Change of tendon related pain on visual analogy scale at 16 weeks | 16 weeks
  Maximal intensity of self-perceived pain in the past 7 days, pain during single-leg declined-squat test
Tendon related dysfunction by questionnaire at baseline | Before intervention
  Victorian Institute of Sport Assessment Questionnaire - Patellar Tendon
Change of tendon related dysfunction by questionnaire at 12 weeks | 12 weeks
  Victorian Institute of Sport Assessment Questionnaire - Patellar Tendon
Change of tendon related dysfunction by questionnaire at 16 weeks | 16 weeks
  Victorian Institute of Sport Assessment Questionnaire - Patellar Tendon

IPD SHARING:
Plan to Share IPD: No
No plan